CLINICAL TRIAL: NCT06655025
Title: The Effects of Dexmedetomidine on Postoperative Cognitive Function and Neuron-Specific Enolase Levels in Open Heart Surgery
Brief Title: The Effects of Dexmedetomidine on Postoperative Cognitive Function in Open Heart Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Salaheldin Ahmed Abdelziz, specialist, Sohag University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Soh-Med-15-10-1MD
Record Dates: First submitted 2024-10-22; First posted 2024-10-23 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Open Heart Sugery; Neuronal Damage
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group B (Dexmedetomidine) (Active Comparator): Dexmedetomidine infusion
  Interventions: Drug: Dexmedetomidine
- Group A (control) (Placebo Comparator): normal saline infusion
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — Dexmedetomidine infusion during open heart surgery

SUMMARY:
To assess the impact of Dexmedetomidine on postoperative cognitive function and serum Neuron Specific Enolase levels as an indicator of neuronal injury in patients undergoing open heart surgery

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes undergoing elective open-heart surgery

Exclusion Criteria:

* Patients with a history of neurological disorders, severe renal or liver dysfunction, or contraindications to Dexmedetomidine as in patients with known QT prolongation, a history of other arrhythmias, symptomatic bradycardia, hypokalemia, or hypomagnesemia, and in patients receiving other drugs known to prolong the QT interval.

Patients with cognitive impairment, mental and psychological illness and chronic alcoholics, drug addicts, abuse of psychotropic substances, illiterate education

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-10-08 (Actual); Primary Completion 2025-10-08 (Estimated); Study Completion 2025-10-08 (Estimated)

PRIMARY OUTCOMES:
postoperative cognitive function | pre- oprerative , Mini-mental state examination (MMSE) will be performed at 1, 3 and 7 days after operation.
  using the Mini-Mental State Examination (MMSE) to evaluate cognitive status

SECONDARY OUTCOMES:
serum Neuron Specific Enolase levels | pre-operative ,post-operative 12 hours
  serum Neuron Specific Enolase levels as an indicator of neuronal injury in patients undergoing open heart surgeries.

OTHER OUTCOMES:
Bispectral index-guided anesthesia depth | BIS will be recorded at induction of anaesthesia (T0), immediately after intubation (T1), when incision will be made (T2), at time of cardiopulmonary bypass (T3) and when operation will be completed (T4).
  To evaluate the effects of Dexmedetomidine on Bispectral index-guided anesthesia depth in patients undergoing open heart surgeries

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided